CLINICAL TRIAL: NCT00159458
Title: Phase II Clinical Trial of Gemcitabine and Oxaliplatin in Recurrent or Metastatic Breast Cancer
Brief Title: Clinical Trial of Gemcitabine and Oxaliplatin in Recurrent or Metastatic Breast Cancer
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Insufficient Accrual
Sponsor: University of Southern California (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 1B-03-1
Record Dates: First submitted 2005-09-08; First posted 2005-09-12 (Estimated); Last update posted 2014-05-22 (Estimated); Status verified 2014-05

CONDITIONS: Recurrent Breast Cancer; Metastastic Breast Cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — Gemcitabine; Oxaliplatin

INTERVENTIONS:
Drug: Gemcitabine and oxaliplatin

SUMMARY:
The purpose of this study is to find out if the combination of gemcitabine and oxaliplatin chemotherapy will be effective in reducing or eliminating the tumor(s) in patients with recurrent or metastatic breast cancer.

Gemcitabine is a chemotherapy drug approved by the U.S. Food and Drug Administration (FDA) for the treatment of pancreatic and lung cancer; oxaliplatin is a chemotherapy drug that is approved by the FDA for the treatment of colon cancer. Neither gemcitabine nor oxaliplatin are approved for the treatment of breast cancer. However, both drugs have been shown to decrease the size of breast cancer tumors.

ELIGIBILITY:
Inclusion Criteria:

* Histologically proven dx of recurrent or metastatic breast cancer
* Must have received at least 1 but not more than 3 prior chemotherapy regimens for recurrent or metastatic breast cancer. Patients who relapse within 12 months of completing adjuvant chemotherapy can only have had up to 2 prior regimens for metastatic disease. Patients who relapse within 12 months of completing adjuvant chemotherapy containing an anthracycline and a taxane, do not require prior chemotherapy for metastatic disease.
* Unidimensionally measurable dz (by RECIST)
* At least 18 yrs of age
* SWOG PS 0-2
* AGC greater than or equal to 1.5; platelets greater than or equal to 100,000; Hgb greater than or equal to 8.0
* Total bilirubin less than or equal to 2 x uln; SGOT and/or SGPT and alk phos up to 2.5 x uln
* Creatinine less than or equal to 2.0
* Fully recovered from acute toxicities secondary to prior tx
* Signed informed consent (including HIPAA authorization)
* Peripheral neuropathy grade 0-1

Exclusion Criteria

* Prior tx with gemcitabine or oxaliplatin. Prior tx with cisplatin or carboplatin allowed if completed >12 mos prior to enrollment.
* Underlying medical, psychiatric, or social conditions that would preclude patient from receiving tx
* Peripheral neuropathy greater than or equal to Gr 2

Exclusion Criteria:

-

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 7 (Actual)
Dates: Start 2003-07; Primary Completion 2006-11 (Actual); Study Completion 2006-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Christy Russell, MD, Principal Investigator — LAC+USC Medical Center
Locations (2):
- United States (2):
  - Norris Comprehensive Cancer Center, Los Angeles, California
  - Premiere Oncology, Santa Monica, California